CLINICAL TRIAL: NCT05115396
Title: Effectiveness of Mirror Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 221021
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror therapy (Experimental): To perform mirror therapy, the participant shall be seated in a chair with a table in front of him/her. On the table there will be a mirror in the sagittal plane between the two upper limbs. The affected hand will be behind the mirror, without visibility, while the hand without symptoms will be reflected laterally in the mirror. Thus, the mirror will reflect the movements of the unaffected side as if these movements were executed with the affected side. During the intervention, participants will be instructed to concentrate on the hand reflected in the mirror.
  During MT, they will perform an exercise protocol based on previous studies and the American College of Sports Medicine guidelines. The duration will be 30 minutes.
  Interventions: Other: Mirror therapy
- Cross-education treatment (Active Comparator): Participants will perform the same exercise protocol with the unaffected hand and without the use of a mirror.
  Interventions: Other: Cross-education treatment

INTERVENTIONS:
Other: Mirror therapy — The patient shall be seated in a chair with a table in front of him/her. On the table there is a mirror in the sagittal plane between the two upper extremities. The affected hand will be behind the mirror, without visibility, while the hand without symptoms will be reflected laterally in the mirror. Thus, the mirror will reflect the movements of the unaffected side as if these movements were executed with the affected side. During the procedure, patients will be instructed to concentrate on the hand reflected in the mirror.
  Arms: Mirror therapy
Other: Cross-education treatment — Participants will perform the same exercise protocol with the unaffected hand and without the use of a mirror.
  Arms: Cross-education treatment

SUMMARY:
Carpal tunnel syndrome (CTS) is the most prevalent entrapment neuropathy. CTS presents with motor and sensory disturbances, including pain, paraesthesia, and numbness in the fingers and hand. Therefore, CTS has a great impact on the activities of daily living.

There are non-surgical treatments that can be effective in people who experience mild or moderate symptoms derived from CTS. Among them, flexor tendon and median nerve sliding exercises may offer an improvement in pain severity and symptoms, strength, wrist joint range, functionality, and quality of life for people with CTS. However, there are few studies on the effectiveness of treatments focused on the mechanisms of neuroplasticity through techniques aimed at rehabilitating different deficits.

Mirror therapy (MT) may be beneficial in musculoskeletal injuries that occur with pain and reduced functionality of a body segment. For example, in people with acute stroke, orthopaedic hand injuries or complex regional pain syndrome type 1. However, its effect has not been studied in patients with CTS in mild or moderate stages.

Thus, the objective of this study is to analyze the effectiveness of MT with conventional CTS exercises in symptoms of median nerve compression, pain, mobility, strength and motor functionality in patients with CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most prevalent entrapment neuropathy. CTS presents with motor and sensory disturbances, including pain, paresthesia, and numbness in the fingers and hand. In addition, since complex movements and tactile sensation of the hand are essential to perform everyday tasks, STC has a great impact on the activities of daily living.

Previuos studies have shown that CTS is not merely a local compression of the median nerve, since associated peripheral and central sensitization phenomena have been verified. In this sense, the decrease in the use of a body segment as a form of protective response to pain, favors the reduction of cortical thickness, affecting the primary motor and somatosensory area. In this way, in patients with CTS it has been described that the modification of the sensory input ends up having an impact on the level of the central nervous system producing different brain plastic changes.

There are non-surgical treatments that can be effective in people who experience mild or moderate symptoms derived from CTS. Among them, flexor tendon and median nerve sliding exercises may offer an improvement in pain severity and symptoms, strength, wrist joint range, functionality, and quality of life for people with CTS. However, there are few studies on the effectiveness of treatments focused on the mechanisms of neuroplasticity through techniques aimed at rehabilitating different deficits.

Mirror therapy (MT), which involves the activation of mirror neurons and contributes to the cortical representation of movement, has been shown to be beneficial in musculoskeletal injuries that occur with pain and reduced functionality of a body segment. Furthermore, it has been shown to be effective in motor recovery of the upper limb in patients with acute stroke, the restoration of joint range and hand function in patients with orthopedic hand injuries, and in the improvement of pain in patients with complex regional pain syndrome type 1.

Similarly, in CTS, the application of MT decreases pain at rest during the night, and improves sensitivity and function in patients undergoing CTS hand surgery. However, its effect has not been studied in patients with CTS in mild or moderate stages where surgical treatment is not urgent or indicated.

Thus, the objective of this study will analyze the effectiveness of MT in combination with conventional exercises compared to conventional exercises on aspects related to symptoms of median nerve compression, pain, joint range, tension strength and motor functionality of the hand in patients with CTS.

Therefore, this study is a randomized clinical trial in which two groups of twenty people in each group will participate, with different interventions:

* Mirror therapy group.
* Cross-education group (without mirror). Participants will receive six-week intervention, 2 supervised sessions per week and 3 unsupervised sessions per week.

Participants will be evaluated in three moments, at baseline, postintervention and one-month-follow-up.

Data analysis will be performed with SPSS statistic program (v26). Normality and homoscedasticity will be analyzed by Shapiro-Wilk t-test and Levene test, respectively. For comparation between groups Bonferroni will be used. If any confusion factor that not meet requirements to be analysed like a covariable exist, ANCOVA will be used. When p<0.0.5 statistical significant differences will be assumed.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age.
* Being diagnosed with CTS
* Unilateral CTS

Exclusion Criteria:

* trauma or surgery on the upper limb within the last two years.
* diagnosis of severe CTS.
* pregnancy.
* atrophy of the tenar muscles.
* local corticosteroid injection or physiotherapy for CTS within the last 3 months.
* peripheral nerve damage.
* entrapment neuropathy at the most proximal levels of the upper limb.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2 minutes
  Visual Analog Scale: 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Symptom severity and functional status | 5 minutes
  Boston Carpal Tunnel Syndrome Questionnaire

SECONDARY OUTCOMES:
Upper limb disability | 5 minutes
  Shortened version of the Disabilities of the Arm, Shoulder, and Hand
Grip and Gripper Strength | 10 minutes
  Dynamometer
Sensitivity | 10 minutes
  Two-point discrimination, and The Semmes-Weinstein monofilament test
Muscle activation | 10 minutes
  BTS FreeEMG electromyograph (wrist flexors, wrist extensors, thumb abductor).
Perception of change after treatment | 2 minutes
  Patient Global Impression of Change Scale: 7-point verbal scale, with the options "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", "very much worse". Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Serra-Añó, Dr, Principal Investigator — Univeristy of Valencia
Locations (2):
- Spain (2):
  - Faculty of Physiotherapy, Valencia, Valencia / València
  - Faculty of Physiotherapy, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thieme H, Morkisch N, Mehrholz J, Pohl M, Behrens J, Borgetto B, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2018 Jul 11;7(7):CD008449. doi: 10.1002/14651858.CD008449.pub3. PMID 29993119
- [Derived] Munoz-Gomez E, Aguilar-Rodriguez M, Molla-Casanova S, Sempere-Rubio N, Ingles M, Serra-Ano P. A randomized controlled trial on the effectiveness of mirror therapy in improving strength, range of movement and muscle activity, in people with carpal tunnel syndrome. J Hand Ther. 2024 Oct-Dec;37(4):534-543. doi: 10.1016/j.jht.2024.02.007. Epub 2024 Mar 7. PMID 38458950